CLINICAL TRIAL: NCT02071134
Title: Registry of Deep Brain Stimulation With the VERCISE™ System: Vercise DBS Registry
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A4010; A4069 (Other: Boston Scientific Corporation U.S. Study)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Parkinson's Disease
Keywords: Deep brain stimulation; Parkinson's disease; Vercise
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Parkinson's disease: Subjects with Parkinson's disease who will receive Vercise DBS for deep brain stimulation.
  Interventions: Device: Deep Brain Stimulation (DBS)

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) — Subjects receiving Deep Brain Stimulation (DBS) for the treatment of their Parkinson's disease symptoms will be offered participation in this registry.
  Other Names: Vercise DBS System; Boston Scientific

SUMMARY:
The purpose of this registry is to compile characteristics of world-wide outcomes for the use of Boston Scientific's commercially available Vercise DBS System in the treatment of Parkinson's disease.

The utilization of Image Guided Programming (IGP), and other commercially available programming features, used as planning tools for the programming of patients with Boston Scientific's Vercise DBS System are also evaluated.

Additionally, the utilization of the DBS Illumina 3D feature that may be used for the programming of patients with Boston Scientific's Vercise DBS Systems is also evaluated.

DETAILED DESCRIPTION:
The purpose of this registry is to compile characteristics of world-wide outcomes for the use of Boston Scientific's commercially available Vercise DBS system in the treatment of Parkinson's disease.

Subjects' improvement in disease symptoms and overall Quality of life will be assessed during the study following DBS and compared with baseline. Additionally, the utilization of Image Guided Programming (IGP) when used as a planning tool for programming of patients is also evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Meets criteria established in locally applicable Vercise System Direction for Use
* At least 18 years old

Key Exclusion Criteria:

* Meets any contraindication in the Vercise System locally applicable Directions for Use

Subjects with significant cognitive or psychiatric impairment may be excluded in the evaluation of GXT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms of Parkinson's disease that are not adequately controlled with medication
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-03-04 (Actual); Primary Completion 2038-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in patient's quality of life (QoL) during the study as compared with baseline | up to 3 years
  Change in quality of life assessments during the study as compared with baseline

OTHER OUTCOMES:
Change in parkinson's disease symptoms as determined by UPDRS scores during the study as compared with baseline | up to 3 years
  Change in patient's motor symptoms as determined by UPDRS during the study as compared with baseline
Change in medication usage during the study as compared with baseline | up to 3 years
Impression of change scores during the study as compared with baseline | 3 years
  Impression of change scores during the study as compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (84):
- United States (28):
  - Neurology and Pain Specialty, Aliso Viejo, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - University of Florida Shands Hospital, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Tallahassee Neurological Clinic, PA, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - St. Luke Regional Medical Center, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Methodist Hospital of Indianapolis, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Louis University Hospital, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - Northwell Health Neuroscience Institute, Great Neck, New York
  - University at Buffalo, Williamsville, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
  - University of Texas Health Medical Arts and Research Center, San Antonio, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Evergreen Health, Kirkland, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Inland Northwest Research, Spokane, Washington
- Fundacion Ineco-Research Facility, Buenos Aires, Argentina
- A.o. LKH Univ.-Kliniken Innsbruck, Innsbruck, Austria
- Belgium (3):
  - AZ Sint-Lucas, Ghent
  - UZ Gasthuisberg, Leuven
  - AZ Delta, Roeselare
- Canada (2):
  - Queen Elizabeth II Health Sciences Center, Halifax
  - Hopital de Enfant-Jesus, Québec
- France (5):
  - CHU Henri Mondor, Créteil
  - Hopital Neurologique Pierre Wertheimer, Lyon
  - CHU La Timone Hospital, Marseille
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - CHRU Hopital Pontchaillou, Rennes
- Germany (11):
  - University Berlin, Charite Virchow Standort, Wedding, Berlin
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinik Eppendorf, Hamburg
  - St. Barbara-Klinik Hamm-Heessen, Hamm
  - Universitätsklinikum Campus Kiel, Kiel
  - Johannes Gutenberg Universitaet Mainz, Mainz
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg
  - Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Universitätsklinikum Würzburg, Würzburg
- Medical School of University PECS, Pécs, Hungary
- Israel (3):
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Italy (7):
  - Villa Margherita, Arcugnano
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Ospedale Dell Angelo, Mestre
  - IRCCS Istituto Ortopedico Galeazzi, Milan
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia
  - Policlinico Universitario Agostino Gemelli, Rome
  - Osp. S. Maria Della Misericordia, Udine
- Poland (3):
  - 10 Military Clinical Hospital Bydgoszcz, Bydgoszcz
  - Podmiot Leczniczy Copernicus Sp. z o.o., Gdansk
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Seoul ASAN Medical Center, Seoul
  - Yonsei University Severance Hospital, Seoul
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital De Bellvitge, Barcelona
  - Centro Especial Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - University Hospital Virgen Arrixaca, Murcia
  - Hospital General De Asturias, Oviedo
- Turkey (Türkiye) (2):
  - Bahcesehir University Hospital Medical Park Goztepe, Istanbul
  - Koc University Hospital, Istanbul
- United Kingdom (8):
  - Southmead Hospital Bristol, Bristol
  - Queen Elizabeth University Hospital, Glasgow
  - The Walton Centre, Liverpool
  - Charing Cross Hospital, London
  - King's College Hospital London, London
  - St. Georges Hospital, London
  - Royal Victoria Infirmary, Newcastle
  - John Radcliffe Hospital, Oxford